CLINICAL TRIAL: NCT02094014
Title: Auditory Masking Effects on Speech Fluency in Aphasia and Apraxia of Speech
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-0503; R03DC011881 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-21 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Apraxia of Speech; Aphasia; Cerebrovascular Accident
Keywords: Perceptual masking; Auditory stimulation; Speech; Language; Verbal Fluency Disorders
MeSH Terms: conditions — Apraxias; Aphasia; Stroke; Speech; Language; Speech Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aphasic/Apraxic Participants: The aphasic/apraxic participant group will include 30 adults who have had strokes affecting their ability to communicate verbally, broadly classified as aphasic and including individuals with and without apraxia of speech (AOS).
  Participants will speak under Masked Auditory Feedback, Altered Auditory Feedback, and Normal Auditory Feedback.
  Interventions: Behavioral: Normal Auditory Feedback; Behavioral: Masked Auditory Feedback; Behavioral: Altered Auditory Feedback
- Neurologically Healthy Participants: The neurologically healthy participant group will include 15 adults with no history of stroke or developmental speech or language disorder.
  Participants will speak under Masked Auditory Feedback, Altered Auditory Feedback, and Normal Auditory Feedback.
  Interventions: Behavioral: Normal Auditory Feedback; Behavioral: Masked Auditory Feedback; Behavioral: Altered Auditory Feedback

INTERVENTIONS:
Behavioral: Normal Auditory Feedback — Participants will produce sentences under normal speaking conditions, able to hear their own speech.
Behavioral: Masked Auditory Feedback — Participants will produce sentences while listening to speech-shaped noise at 85 decibels (sound pressure level) to mask ability to hear their own speech.
  Other Names: Masking Noise
Behavioral: Altered Auditory Feedback — Participants will produce sentences while listening to their speech shifted up one octave and delayed.
  Other Names: Delayed and pitch-shifted feedback

SUMMARY:
Impaired speech production is a major obstacle to full participation in life roles by stroke survivors with aphasia and apraxia of speech. The proposed study will demonstrate the short-term effects of auditory masking on speech disfluencies and identify individual factors that predict a positive response, enabling future work to develop auditory masking as a treatment adjuvant targeting long-term improvement in speech. Providing an additional treatment option for adults with aphasia and apraxia of speech will have the clear benefit of improving quality of life and allowing individuals to participate more actively in their health care decisions through improved communication.

DETAILED DESCRIPTION:
The objective of this research is to test the short-term effects of listening to noise (i.e. auditory feedback masking) on speech fluency in stroke survivors with aphasia and apraxia of speech. People with nonfluent types of aphasia frequently have apraxia of speech, which affects the motor programming of speech movements, causing distortions, slow rate, and speech disfluencies that impede the forward flow of communication. Speaking while listening to noise (e.g. auditory masking) is known to reduce disfluencies and increase speech rate in people who stutter. This method has been tested in people with aphasia, resulting in positive effects on speech production for a subset of those tested. The investigators contend that individuals who have apraxia of speech in addition to aphasia are most likely to benefit from auditory masking, but most previous studies did not test participants for apraxia of speech. In addition, though masking is most likely to affect speech disfluencies, previous studies did not measures disfluencies. The proposed work has two specific aims. Aim 1 will determine the short-term effect of auditory masking, provided on a single day, on speech fluency in stroke survivors with aphasia and apraxia of speech. Aim 2 will identify individual factors that predict a positive response, including presence of apraxia of speech, lesion characteristics, and type of aphasia (e.g. Broca's, Wernicke's). Voxel-based lesion analysis techniques will be used to determine sites of lesion associated with positive and negative response to auditory masking. Completion of this study will remove barriers to studying auditory masking as a technique for clinical intervention, but also as a research tool for behavioral neuroscientists probing the speech motor control system in speakers with aphasia and apraxia of speech.

ELIGIBILITY:
Inclusion Criteria for Aphasic/Apraxic Participants:

* Single left-hemisphere cerebrovascular accident
* Speech errors are present, but participant is able to produce approximations of words or sentences by reading or repetition; < 90% and > 10% on Chapel Hill Multilingual Intelligibility Test (Haley, 2011)
* Right-handed prior to stroke by report
* Normal visual attention, acuity, and color vision
* Pure-tone threshold <= 40 decibels in at least one ear

Exclusion Criteria for Aphasic/Apraxic Participants:

* Predominating disorders of cognition or hearing (e.g. dementia, hearing impairment).
* Presence of degenerative neurological illness (e.g. Parkinson's disease, amyotrophic lateral sclerosis, primary progressive aphasia).

Inclusion Criteria for Neurologically Healthy Participants:

* Matched in age and sex to a participant with aphasia
* score of 90% or higher on the single-word intelligibility test
* Right-handed prior to stroke by report
* Normal visual attention, acuity, and color vision
* Pure-tone threshold <= 40 decibels in at least one ear

Exclusion Criteria for Neurologically Healthy Participants:

* History of stroke
* History of developmental speech or language disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with aphasia (PWA) will be referred from existing referral sources (e.g. UNC Stroke registry, Triangle Aphasia Project), clinicians in the community, and the Carolina Data Warehouse for Health.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Disfluency duration change with masking noise | 1 day of the study
  Measured disfluency duration in sentences produced while listening to masking noise compared to speaking in quiet without noise.

SECONDARY OUTCOMES:
Speech rate change with masking noise | 1 day of the study
  Measured syllables per second in sentences produced while listening to masking noise compared to speaking in quiet without noise.
Speech sound accuracy change with masking noise | 1 day of the study
  Measured speech sound accuracy in sentences produced while listening to masking noise compared to speaking in quiet without noise.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Jacks, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States